CLINICAL TRIAL: NCT06076408
Title: Effects of Sustained Natural Apophyseal Glides With and Without Pilates on Pain, Range of Motion and Disability in Patients With Lumbar Disc Bulge
Brief Title: Effects of SNAGS With and Without Pilates in Lumbar Disc Bulge Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/0165Ammar Javed
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Lumbar Disc Herniation; Lumbar Radiculopathy
Keywords: disability; lumbar radiculopathy; low back pain; endurance
MeSH Terms: conditions — Intervertebral Disc Displacement; Radiculopathy; Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SNAGS with Pilates (Experimental): Sustained Natural Apophyseal glides and Pilates Exercises
  Interventions: Other: SNAGS with Pilates
- SNAGS (Active Comparator): Sustained Natural Apophyseal glides
  Interventions: Other: SNAGS

INTERVENTIONS:
Other: SNAGS with Pilates — Patients will Receive Sustained Natural Apophyseal glides and Pilates Technique. Pilates Exercises focusses on five main areas (breath control, pelvic lumbar region, chest, shoulder positioning, head and neck positioning) a special session was organized for each patient
  Arms: SNAGS with Pilates
Other: SNAGS — Patients will Receive Sustained Natural Apophyseal glides
  Arms: SNAGS

SUMMARY:
The aim of this study is to compare the effects of Sustained Natural Apophyseal Glides with and without Pilates on pain, range of motion and disability in patients with lumbar Disc Bulge.

DETAILED DESCRIPTION:
Lumbar disc disease may occur when a disc in the low back area of the spine bulges or herniates between the bony areas of the spine. Lumbar disk disease causes lower back pain and leg pain and weakness that is made worse by movement and activity. Lumbar disc bulge is typically managed through a multidimensional approach that integrates various therapeutic techniques aimed at reducing symptoms and enhancing functional outcomes. The use of SNAGs has been shown to produce positive results such as decreased pain levels and increased mobility in previous studies. Overall physical conditioning can be improved by using a holistic approach that consists of controlled movements combined with breathing techniques and mindfulness. In order to treat lumbar disc bulge patients more effectively, it is important to understand how use and efficacy differ when applying SNAGs alone versus together with Pilates. Delving into how combining SNAGs and Pilates affects lumbar disc bulge patients contributes to an expanding body of proof advocating for a multimodal treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient of both gender under the age of 40-60 year.
* Unilateral radiating pain through the course of sciatic nerve
* a duration of pain of at least 3 months
* Restricted lumbar range of motion.
* Subjects who can understand the instructions and are willing to participate in the study
* Positive slump test with positive pain location and positive pain descriptors.
* Passive Lumbar Extension If the patient experiences severe low back pain or if there is a feeling of heaviness on the lower back or a feeling as though the lower back were about to 'come off' the test is considered positive.
* Straight Leg Raise SLR test positive when it evokes radiating pain along the course of the sciatic nerve and below the knee between 30 and 70 degrees of hip flexion

Exclusion Criteria:

* History of trauma, dislocation and subluxation of lower extremity.
* Rheumatoid Arthritis
* Systemic diseases such as blood coagulation disorders, chronic pain syndrome, cancer, allergies fibromyalgia, systemic lupus erythematous, and psoriatic arthritis.
* Lumbar spine surgery patients.
* Malignancy
* neurologic disorders (e.g., trigeminal neuralgia or occipital neuralgia)
* clinical diagnosis of lumbar bilateral radiculopathy or myelopathy
* history of previous physical therapy intervention for the lumbar region in last 6 months

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 3 weeks
  NPRS scale can be used to quantify pain intensity levels. The 11-point scale ranges from '0' for the least amount of pain "no pain" to '10' for the most extreme levels of pain "pain as severe as you can imagine". It is convenient to use NPRS for patients. Its score ranges between 0-10. "change will be measured from baseline to 3 weeks"
Modified Oswestry Disability Index | 3 weeks
  The ODI is a disease specific disability measure is used to establish measure a level of disability stage of patients' acuity status and monitor change over time. The final score ranges from 0-100. A score of 0-20 reflects minimal disability, 21-40 moderate disability, 41-60 severe disability, 61-80 crippled, and 81-100 bed-bound. "Change will be measured from baseline to 3 weeks"
Lumbar ROM by inclinometer | 3 weeks
  Inclinometer is used to measure the range of motion on Lumbar spine. "Change in ROM will be measured from baseline to 3 weeks".

CONTACTS AND LOCATIONS:
Overall Officials: Faiza Ashraf, TDPT, Principal Investigator — Riphah International University; Ammar Javed, MS OMPT*, Principal Investigator — Riphah International University
Locations (1):
- Bakhtawar Amin Hospital Multan, Multan, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No